CLINICAL TRIAL: NCT04903496
Title: Characteristics, Treatment, and Economic Burden of Disease of Chinese Diabetic/Non-diabetic Patients With/Without Established Cardiovascular Disease, Chronic Kidney Disease, or at High Cardiovascular Risk
Brief Title: Clinical Characteristics and Disease Burden of Diabetic Patients Based on Tianjin Regional Database
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Chengdu Big Data Association (Industry)
Responsible Party: Sponsor
Other Study IDs: 1245-0203
Record Dates: First submitted 2021-05-25; First posted 2021-05-26 (Actual); Results first posted 2024-11-12 (Actual); Last update posted 2024-11-12 (Actual); Status verified 2024-09

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- In- and outpatients: diabetic with risk factors (RF) [Arm A]: In- and outpatients with diagnosis of diabetes, and with diagnosis of risk factors cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD) or at high cardiovascular (CV) risk identified in the Tianjin regional medical database.
- In- and outpatients: diabetic without RF [Arm B]: In- and outpatients with diagnosis of diabetes, but not with diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database.
- In- and outpatients: non-diabetic with RF [Arm C]: In- and outpatients without diabetes but with diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database.
- In- and outpatients: non-diabetic without RF [Arm D]: In- and outpatients without diabetes and without diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database.

SUMMARY:
The study aims to investigate the clinical characteristics, treatment, and economic burden of disease of Chinese diabetic/non-diabetic patients with/without established cardiovascular disease (CVD), chronic kidney disease (CKD), or at high cardiovascular risk, including:

* Primary objectives: describe the proportion of Chinese diabetic/non-diabetic patients with established cardiovascular disease, CKD, or at high cardiovascular risk including hypertension and hyperlipidemia
* Secondary objectives: describe the demographic characteristics of the last visit for all patients, and the demographic characteristics of inpatients over time; investigate the clinical characteristic for all patients

ELIGIBILITY:
Inclusion Criteria:

* Patients in the Tianjin regional database from 01/01/2015 to 31/12/2019
* Group A: patients with diagnosis of diabetes, and with diagnosis of cardiovascular disease, heart failure, chronic kidney disease or at high cardiovascular risk
* Group B: patients with diagnosis of diabetes, but not with diagnosis of cardiovascular disease, heart failure, chronic kidney disease or at high cardiovascular risk
* Group C: patients with diagnosis of cardiovascular disease, heart failure, chronic kidney disease or at high cardiovascular risk, but not with diagnosis of diabetes
* Group D: patients without diagnosis of cardiovascular disease, heart failure, chronic kidney disease or at high cardiovascular risk, and without diagnosis of diabetes. We will randomly select a group of non-diabetic patients without any of the above diseases by matching on age and gender

Definition of diabetes, cardiovascular disease, chronic kidney disease and high cardiovascular risk:

* Diabetes: patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of diabetes (the first diagnosis will be the index diagnosis, and the time interval between diagnoses is not restricted) (International classification of disease (ICD)-10 E10-E14);
* Cardiovascular disease: patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of ischemic heart diseases (the first diagnosis will be the index diagnosis, and the time interval between diagnoses is not restricted) (ICD-10 I20~I25); or patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of cerebrovascular diseases (the first diagnosis will be the index diagnosis, and the time interval between diagnoses is not restricted) (ICD-10 I60~I69); or patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of ischemic peripheral artery disease (the first diagnosis will be the index diagnosis, and the time interval between diagnoses is not restricted) (ICD-10 E10.501, E11.603, E14.501, E14.606, E14.503, I73.9, I99.03, I99.04);
* Heart failure: patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of heart failure (the first diagnosis will be the index diagnosis, and the time interval between diagnoses is not restricted) (ICD-10 I50);
* Chronic kidney disease (CKD): inpatients with at least once 1 discharged diagnosis CKD (ICD-10 N18), or inpatients with the last estimated glomerular filtration rate (eGFR, calculated by Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation) <60 mL/min/1.73 m2 or prescription of dialysis, but not with the diagnosis of acute kidney injury (ICD-10 N17); or outpatients with at least 2 diagnosis of CKD (the first diagnosis will be the index diagnosis, and the time interval between diagnoses is not restricted) or with two consecutive eGFR (calculated by CKD-EPI equation) <60 mL/min/1.73 m2 by 90 days or more;
* High cardiovascular risk: patients with at least 1 discharged diagnosis or 2 outpatient diagnosis of hypertension (the first diagnosis will be the index diagnosis, and the time interval between diagnoses is not restricted) (ICD-10 I10~I15); or at least 1 discharged diagnosis or 2 outpatient diagnosis of hyperlipidemia (ICD-10 E78.001-E78.003, E78.101, E78.203, E78.301-E78.304, E78.306, E78.401, E78.501, E78.902);

Exclusion Criteria:

* Patients with non-Chinese nationalities
* Duplicated storage (records with same inpatient code)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diabetic/non-diabetic patients with/without established cardiovascular disease, chronic kidney disease, or at high cardiovascular risk.
Sampling Method: Non-Probability Sample
Enrollment: 1233162 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-06-24 (Actual); Study Completion 2022-06-24 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Chengdu Big Data Association, Chengdu, China

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This observational, cross-sectional study, based on routinely collected data captured in the regional, electronic, data-linking Tianjin medical database between 01/01/2015 and 31/12/2019 aimed to investigate the clinical characteristics, treatment, and economic burden of disease of Chinese diabetic/non-diabetic patients with/without established cardiovascular disease, chronic kidney disease, or high cardiovascular risk.
Pre-assignment Details: Only participants that met all inclusion and none of the exclusion criteria were included. Participants with at least 1 diagnosis record and baseline information (birth date and sex) were identified in the Tianjin regional medical database between 01/01/2015 to 31/12/2019 and allocated in 4 (A,B,C, and D) arms. The 4 arms were mutually exclusive in each year (2015, 2017, and 2019) but not across years.
Period: Study Period 2015
Arm/Group | In- and Outpatients: Diabetic With Risk Factors (RF) [Arm A] | In- and Outpatients: Diabetic Without RF [Arm B] | In- and Outpatients: Non-diabetic With RF [Arm C] | In- and Outpatients: Non-diabetic Without RF [Arm D]
Started | 166056 | 113787 | 66525 | 51640
Completed | 166056 | 113787 | 66525 | 51640
Not Completed | 0 | 0 | 0 | 0
Period: Study Period 2017
Arm/Group | In- and Outpatients: Diabetic With Risk Factors (RF) [Arm A] | In- and Outpatients: Diabetic Without RF [Arm B] | In- and Outpatients: Non-diabetic With RF [Arm C] | In- and Outpatients: Non-diabetic Without RF [Arm D]
Started | 379826 | 188681 | 144484 | 123839
Completed | 379826 | 188681 | 144484 | 123839
Not Completed | 0 | 0 | 0 | 0
Period: Study Period 2019
Arm/Group | In- and Outpatients: Diabetic With Risk Factors (RF) [Arm A] | In- and Outpatients: Diabetic Without RF [Arm B] | In- and Outpatients: Non-diabetic With RF [Arm C] | In- and Outpatients: Non-diabetic Without RF [Arm D]
Started | 576973 | 253012 | 198099 | 205078
Completed | 576973 | 253012 | 198099 | 205078
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Number of participants with at least one recorded International Classification of Disease (ICD) code diagnosis in the Tianjin regional database, Chinese nationality, and baseline information (birth date and sex) in 2015, 2017, and 2019.
Groups:
- All in- and Outpatients [Arm A, B, C, D Together] in 2015, 2017, and 2019: All in- and outpatients with and without diagnosis of diabetes and with and without established risk factors cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD), or at high cardiovascular (CV) risk.
Arm/Group | All in- and Outpatients [Arm A, B, C, D Together] in 2015, 2017, and 2019
Number analyzed (Participants) | 1233162
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: As per protocol baseline characteristics were calculated by year over all individual participants considering only participants with available data at their last visit.
  Years
    All in- and outpatients in 2015: number analyzed (Participants) | 398008
    All in- and outpatients in 2015 | 60.1 (12.9)
    All in- and outpatients in 2017: number analyzed (Participants) | 580958
    All in- and outpatients in 2017 | 59.3 (13.1)
    All in- and outpatients in 2019: number analyzed (Participants) | 680438
    All in- and outpatients in 2019 | 58.9 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: As per protocol baseline characteristics were calculated by year over all individual participants considering only participants with available data at their last visit.
  Participants
    All in- and outpatients in 2015: number analyzed (Participants) | 398008
    All in- and outpatients in 2015: Female | 195654
    All in- and outpatients in 2015: Male | 202354
    All in- and outpatients in 2017: number analyzed (Participants) | 580958
    All in- and outpatients in 2017: Female | 287609
    All in- and outpatients in 2017: Male | 293349
    All in- and outpatients in 2019: number analyzed (Participants) | 680438
    All in- and outpatients in 2019: Female | 335474
    All in- and outpatients in 2019: Male | 344964
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Established Cardiovascular Disease, or Chronic Kidney Disease, or High Cardiovascular Risk
Description: Number of participants with established cardiovascular disease (CVD), chronic kidney disease (CKD), and/or high cardiovascular (CV) risk was calculated as (100%* Number of patients with labels of interested diseases from 2015 to the given year)/ (Number of diabetic or non-diabetic patients from 2015 to the given year).
  To compare diabetic with non-diabetic patients within a year and across years
  * the arms with diabetic in- and outpatients [Arm A and B together] were combined
  * the arms with non-diabetic in- and outpatients [Arm C and D together] were combined by year.
  Patients with risk factors were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: up to 5 years (2015 up to 2019)
Population: In- and outpatients in 2015, 2017, and 2019 with and without diabetes and with and without diagnosis of risk factors CVD, HF, CKD, and high CV risk. For this outcome, groups were combined as per protocol to 'Diabetic Patients [Arm A and B]' and 'Non-Diabetic Patients [Arm C and D]'. Arms were not mutually exclusive. Only patients with available data were included in this analysis.
Measure: Count of Participants; unit: Participants
Groups:
- Diabetic In-and Outpatients in 2015 [Arm A and B]: In-and outpatients with diabetes, and with or without diagnosis of risk factors cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD), or high cardiovascular (CV) risk recorded in the Tianjin regional database in 2015.
- Non-diabetic In-and Outpatients in 2015 [Arm C and D]: In-and outpatients without diabetes, and with or without diagnosis of risk factors CVD, HF, CKD, or high CV risk recorded in the Tianjin regional database in 2015.
- Diabetic In-and Outpatients in 2017 [Arm A and B]: In-and outpatients with diabetes, and with or without diagnosis of risk factors CVD, HF, CKD, or high CV risk and were recorded in the Tianjin regional database in 2017.
- Non-diabetic In-and Outpatients in 2017 [Arm C and D]: In-and outpatients without diabetes, and with or without diagnosis of risk factors CVD, HF, CKD, or high CV risk and were recorded in the Tianjin regional database in 2017.
- Diabetic In-and Outpatients in 2019 [Arm A and B]: In-and outpatients with diabetes, and with or without diagnosis of risk factors CVD, HF, CKD, or high CV risk and were recorded in the Tianjin regional database in 2019.
- Non-diabetic In-and Outpatients in 2019 [Arm C and D]: In-and outpatients without diabetes, and with or without diagnosis of risk factors CVD, HF, CKD, or high CV risk and were recorded in the Tianjin regional database in 2019.
Arm/Group | Diabetic In-and Outpatients in 2015 [Arm A and B] | Non-diabetic In-and Outpatients in 2015 [Arm C and D] | Diabetic In-and Outpatients in 2017 [Arm A and B] | Non-diabetic In-and Outpatients in 2017 [Arm C and D] | Diabetic In-and Outpatients in 2019 [Arm A and B] | Non-diabetic In-and Outpatients in 2019 [Arm C and D]
Number analyzed (Participants) | 279843 | 118165 | 568507 | 268323 | 829985 | 403177
Participants
  With cardiovascular disease | 127726 | 43819 | 295882 | 99128 | 448063 | 138069
  With chronic kidney disease | 16143 | 2465 | 47900 | 7059 | 89826 | 13012
  High cardiovascular risk | 113261 | 52628 | 293826 | 115692 | 473348 | 159502

2. Secondary Outcome: Mean Age of Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2015
Description: The mean age was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2015, up to 1 day
Population: In- and outpatients in 2015 with and without diabetes and with and without diagnosis of risk factors CVD, HF, CKD, and high CV risk. For this outcome, inpatients results [Arm A, B, C, D] are reported separately per arm and in- and outpatients results [All in-and outpatients] are reported over all in- and outpatients and over all arms in 2015. Only patients with available data for this outcome were included in this analysis.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015: Inpatients with diabetes, and with diagnosis of risk factors cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD) or at high cardiovascular (CV) risk identified in the Tianjin regional medical database in 2015.
- Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015: Inpatients with diabetes, and without diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2015.
- Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2015: Inpatients without diabetes, and with diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2015.
- Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015: Inpatients without diabetes, and without diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2015.
- All in- and Outpatients in 2015 = Total in 2015: This arm combines all inpatients from arms A, B, C, and D, as well as all outpatients identified in the Tianjin regional medical database in 2015. This arm takes into account all cases of both inpatients and outpatients, with and without diabetes, and with or without a diagnosis of risk factors for cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD), or those at high cardiovascular risk, as identified in the Tianjin regional medical database in 2015.
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 84600 | 14322 | 21682 | 6573 | 398008
Years | 64.1 (12.0) | 49.7 (16.0) | 64.8 (13.3) | 61.9 (12.6) | 60.1 (12.9)

3. Secondary Outcome: Mean Age of Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2017
Description: The mean age was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2017, up to 1 day
Population: In- and outpatients in 2017 with and without diabetes and with and without diagnosis of risk factors CVD, HF, CKD, and high CV risk. For this outcome, inpatients results [Arm A, B, C, D] are reported separately per arm and in- and outpatients results [All in-and outpatients] are reported over all in- and outpatients and over all arms in 2017. Only patients with available data for this outcome were included in this analysis.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017: Inpatients with diabetes, and with diagnosis of risk factors cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD) or at high cardiovascular (CV) risk identified in the Tianjin regional medical database in 2017.
- Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017: Inpatients with diabetes, and without diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2017.
- Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017: Inpatients without diabetes, and with diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2017.
- Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017: Inpatients without diabetes, and without diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2017.
- All in- and Outpatients in 2017 = Total in 2017: This arm combines all inpatients from arms A, B, C, and D, as well as all outpatients identified in the Tianjin regional medical database in 2017. This arm takes into account all cases of both inpatients and outpatients, with and without diabetes, and with or without a diagnosis of risk factors for cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD), or those at high cardiovascular risk, as identified in the Tianjin regional medical database in 2017.
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 116799 | 22212 | 26955 | 8908 | 580958
Years | 63.0 (12.3) | 44.2 (16.5) | 62.7 (13.8) | 62.1 (12.7) | 59.3 (13.1)

4. Secondary Outcome: Mean Age of Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2019
Description: The mean age was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2019, up to 1 day
Population: In- and outpatients in 2019 with and without diabetes and with and without diagnosis of risk factors CVD, HF, CKD, and high CV risk. For this outcome, inpatients results [Arm A, B, C, D] are reported separately per arm and in- and outpatients results [All in-and outpatients] are reported over all in- and outpatients and over all arms in 2019. Only patients with available data for this outcome were included in this analysis.
Measure: Mean (Standard Deviation); unit: Years
Groups:
- Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019: Inpatients with diabetes, and with diagnosis of risk factors cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD) or at high cardiovascular (CV) risk identified in the Tianjin regional medical database in 2019.
- Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019: Inpatients with diabetes, and without diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2019.
- Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019: Inpatients without diabetes, and with diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2019.
- Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019: Inpatients without diabetes, and without diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2019.
- All in- and Outpatients in 2019 = Total in 2019: This arm combines all inpatients from arms A, B, C, and D, as well as all outpatients identified in the Tianjin regional medical database in 2019. This arm takes into account all cases of both inpatients and outpatients, with and without diabetes, and with or without a diagnosis of risk factors for cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD), or those at high cardiovascular risk, as identified in the Tianjin regional medical database in 2019.
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 139535 | 21549 | 28868 | 9012 | 680438
Years | 61.8 (11.4) | 46.3 (16.2) | 63.0 (12.8) | 62.5 (12.1) | 58.9 (12.9)

5. Secondary Outcome: Number of Female and Male Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2015
Description: The number of female and male was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2015, up to 1 day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Groups:
- Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015: Inpatients without diabetes, and with diagnosis of risk factors CVD, HF, CKD or at high CV risk identified in the Tianjin regional medical database in 2015.
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 84600 | 14322 | 21682 | 6573 | 398008
Participants
  Female | 42775 | 7683 | 11709 | 2761 | 195654
  Male | 41825 | 6639 | 9973 | 3812 | 202354

6. Secondary Outcome: Number of Female and Male Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2017
Description: The number of female and male was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2017, up to 1 day
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 116799 | 22212 | 26955 | 8908 | 580958
Participants
  Female | 54221 | 14543 | 13939 | 3789 | 287609
  Male | 62578 | 7669 | 13016 | 5119 | 293349

7. Secondary Outcome: Number of Female and Male Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2019
Description: The number of female and male was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2019, up to 1 day
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 139535 | 21549 | 28868 | 9012 | 680438
Participants
  Female | 63480 | 14309 | 14894 | 3865 | 335474
  Male | 76055 | 7240 | 13974 | 5147 | 344964

8. Secondary Outcome: Number of Inpatients and All Participants (In-and Outpatients) With Insurance Payment at Their Last Visit in 2015
Description: The number of participants with insurance payment was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2015, up to 1 day
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 84600 | 14322 | 21682 | 6573 | 398008
Participants | 57950 | 8489 | 13797 | 3760 | 340909

9. Secondary Outcome: Number of Inpatients and All Participants (In-and Outpatients) With Insurance Payment at Their Last Visit in 2017
Description: The number of participants with insurance payment was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2017, up to 1 day
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 116799 | 22212 | 26955 | 8908 | 580958
Participants | 77385 | 12792 | 16484 | 4467 | 482628

10. Secondary Outcome: Number of Inpatients and All Participants (In-and Outpatients) With Insurance Payment at Their Last Visit in 2019
Description: The number of participants with insurance payment was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2019, up to 1 day
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 139535 | 21549 | 28868 | 9012 | 680438
Participants | 94453 | 13508 | 18762 | 5167 | 543328

11. Secondary Outcome: Number of Inpatients and All Participants (In-and Outpatients) by Discharge Department at Their Last Visit in 2015
Description: The number of participants in a particular discharge department was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses and records in multiple discharge departments simultaneously. Thus, one participant could potentially occur more than once per arm.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2015, up to 1 day
Population: In- and outpatients in 2015 with and without diabetes and with and without diagnosis of risk factors CVD, HF, CKD, and high CV risk. Inpatients results [Arm A, B, C, D] are reported separately per arm, in- and outpatients results [All in-and outpatients] are reported over all in- and outpatients and over all arms in 2015. Only patients with available data were included in this analysis. Patients could have records in multiple departments or could not be classified to any given department.
Measure: Number; unit: Participants
Groups:
- Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015: Inpatients with diagnosis of diabetes, and with diagnosis of risk factors cardiovascular disease (CVD), heart failure (HF), chronic kidney disease (CKD) or at high cardiovascular (CV) risk identified in the Tianjin regional medical database in 2015.
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 84515 | 14304 | 21619 | 6573 | 397835
Participants
  Department of Pediatric | 210 | 19 | 66 | 2 | 417
  Department of Obstetrics and Gynecology | 933 | 3296 | 420 | 248 | 6897
  Emergency Department | 0 | 0 | 0 | 0 | 7553
  Department of Mental Health | 11 | 5 | 1 | 0 | 876
  Department of Stomatology | 97 | 64 | 42 | 62 | 3719
  Department of Internal Medicine | 58775 | 4829 | 14031 | 1513 | 236691
  Other departments | 3209 | 1221 | 680 | 568 | 85650
  Department of Surgery | 13877 | 4686 | 4890 | 4116 | 39274
  Medical Technical Departments | 19 | 21 | 2 | 4 | 2185
  Department of Integrated Traditional Chinese and Western Medicine | 2769 | 250 | 461 | 21 | 19206
  Department of Critical Care Medicine | 2467 | 80 | 678 | 39 | 2331

12. Secondary Outcome: Number of Inpatients and All Participants (In-and Outpatients) by Discharge Department at Their Last Visit in 2017
Description: The number of participants in a particular discharge department was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses and records in multiple discharge departments simultaneously. Thus, one participant could potentially occur more than once per arm. Thus, one participant could potentially occur more than once per arm.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2017, up to 1 day
Population: In- and outpatients in 2017 with and without diabetes and with and without diagnosis of risk factors CVD, HF, CKD, and high CV risk. Inpatients results [Arm A, B, C, D] are reported separately per arm, in- and outpatients results [All in-and outpatients] are reported over all in- and outpatients and over all arms in 2017. Only patients with available data were included in this analysis. Patients could have records in multiple departments or could not be classified to any given department.
Measure: Number; unit: Participants
Groups:
- Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017: This group includes all inpatients that were of Chinese nationality, without ICD code diagnosis of diabetes, and without ICD code diagnosis of established CVD, CKD, or high CV risk and were recorded in the Tianjin regional database in 2017.
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 116675 | 22189 | 26915 | 8908 | 580764
Participants
  Department of Pediatric | 35 | 136 | 13 | 5 | 422
  Department of Obstetrics and Gynecology | 2071 | 9474 | 659 | 385 | 15681
  Emergency Department | 671 | 66 | 180 | 14 | 14294
  Department of Mental Health | 1 | 0 | 0 | 2 | 1523
  Department of Stomatology | 169 | 83 | 43 | 85 | 3285
  Department of Internal Medicine | 78467 | 5348 | 16959 | 2046 | 358282
  Other departments | 3197 | 1012 | 751 | 630 | 111242
  Department of Surgery | 21583 | 5542 | 6654 | 5571 | 57355
  Medical Technical Departments | 181 | 48 | 59 | 36 | 2180
  Department of Integrated Traditional Chinese and Western Medicine | 3996 | 310 | 571 | 91 | 24076
  Department of Critical Care Medicine | 2623 | 112 | 664 | 43 | 2595

13. Secondary Outcome: Number of Inpatients and All Participants (In-and Outpatients) by Discharge Department at Their Last Visit in 2019
Description: The number of participants in a particular discharge department was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses and records in multiple discharge departments simultaneously. Thus, one participant could potentially occur more than once per arm.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2019, up to 1 day
Population: In- and outpatients in 2019 with and without diabetes and with and without diagnosis of risk factors CVD, HF, CKD, and high CV risk. Inpatients results [Arm A, B, C, D] are reported separately per arm, in- and outpatients results [All in-and outpatients] are reported over all in- and outpatients and over all arms in 2019. Only patients with available data were included in this analysis. Patients could have records in multiple departments or could not be classified to any given department.
Measure: Number; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 138983 | 21549 | 28742 | 9012 | 679661
Participants
  Department of Pediatric | 50 | 229 | 13 | 8 | 704
  Department of Obstetrics and Gynecology | 2428 | 9362 | 686 | 319 | 16314
  Emergency Department | 723 | 92 | 130 | 13 | 18809
  Department of Mental Health | 9 | 0 | 1 | 0 | 1877
  Department of Stomatology | 183 | 70 | 54 | 73 | 3546
  Department of Internal Medicine | 90932 | 4638 | 17288 | 1916 | 408554
  Other departments | 4396 | 1072 | 879 | 688 | 131976
  Department of Surgery | 28099 | 5411 | 7790 | 5864 | 78429
  Medical Technical Departments | 189 | 49 | 72 | 35 | 3325
  Department of Integrated Traditional Chinese and Western Medicine | 4624 | 298 | 665 | 64 | 28303
  Department of Critical Care Medicine | 3081 | 78 | 629 | 30 | 2938

14. Secondary Outcome: Number of Deaths in Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2015
Description: The number of participants who were diagnosed as dead in 2015 was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: On the last visit (1 day) in 2015 data was retrospectively assessed for the last 12 months in 2015.
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 84600 | 14322 | 21682 | 6573 | 398008
Participants | 303 | 18 | 94 | 15 | 430

15. Secondary Outcome: Number of Deaths in Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2017
Description: The number of participants who were diagnosed as dead in 2017 was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: On the last visit (1 day) in 2017 data was retrospectively assessed for the last 12 months in 2017.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 116799 | 22121 | 26955 | 8908 | 580958
Participants | 504 | 29 | 141 | 30 | 704

16. Secondary Outcome: Number of Deaths in Inpatients and All Participants (In-and Outpatients) at Their Last Visit in 2019
Description: The number of participants who were diagnosed as dead in 2019 was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: On the last visit (1 day) in 2019 data was retrospectively assessed for the last 12 months in 2019.
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 139535 | 21549 | 28868 | 9012 | 680438
Participants | 225 | 8 | 41 | 20 | 294

17. Secondary Outcome: The Value of Glycated Hemoglobin (HbA1c) in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2015
Description: The value of glycated hemoglobin (HbA1c) was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2015, up to 1 day
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Percentage of glycated hemoglobin
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 9217 | 1517 | 738 | 2 | 11900
Percentage of glycated hemoglobin | 7.8 [6.9 to 9.3] | 9.2 [7.4 to 11.0] | 5.7 [5.4 to 6.0] | 5.4 [5.3 to 5.4] | 6.9 [6.1 to 8.1]

18. Secondary Outcome: The Value of Glycated Hemoglobin (HbA1c) in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2017
Description: The value of glycated hemoglobin (HbA1c) was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2017, up to 1 day
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Percentage of glycated hemoglobin
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 19404 | 3578 | 1596 | 22 | 26183
Percentage of glycated hemoglobin | 7.6 [6.6 to 9.0] | 7.8 [6.2 to 10.0] | 5.8 [5.6 to 6.2] | 5.8 [5.4 to 6.1] | 7.2 [6.6 to 8.4]

19. Secondary Outcome: The Value of Glycated Hemoglobin (HbA1c) in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2019
Description: The value of glycated hemoglobin (HbA1c) was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2019, up to 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Percentage of glycated hemoglobin
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 50815 | 5093 | 2927 | 49 | 72815
Percentage of glycated hemoglobin | 7.7 [6.8 to 9.1] | 7.3 [6.0 to 9.3] | 5.8 [5.5 to 6.1] | 5.4 [5.1 to 5.7] | 7.1 [6.4 to 8.1]

20. Secondary Outcome: Concentration of Random Blood Glucose in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2015
Description: The concentration (Millimole per liter (mmol/L)) of random blood glucose was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2015, up to 1 day
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Millimole per liter (mmol/L)
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 11534 | 2909 | 3153 | 21 | 19066
Millimole per liter (mmol/L) | 8.3 [6.2 to 12.1] | 8.3 [6.2 to 12.6] | 5.3 [4.7 to 6.1] | 8.5 [6.3 to 10.8] | 8.3 [6.5 to 10.9]

21. Secondary Outcome: Concentration of Random Blood Glucose in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2017
Description: The concentration (Millimole per liter (mmol/L)) of random blood glucose was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2017, up to 1 day
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Millimole per liter (mmol/L)
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 24077 | 6389 | 6065 | 13 | 41511
Millimole per liter (mmol/L) | 9.4 [7.0 to 12.4] | 8.8 [6.5 to 11.3] | 5.3 [4.7 to 6.2] | 7.2 [5.9 to 10.5] | 8.5 [6.8 to 11.3]

22. Secondary Outcome: Concentration of Random Blood Glucose in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2019
Description: The concentration (Millimole per liter (mmol/L)) of random blood glucose was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2019, up to 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Millimole per liter (mmol/L)
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 60298 | 9690 | 12107 | 34 | 119972
Millimole per liter (mmol/L) | 9.0 [6.8 to 12.1] | 7.7 [5.7 to 11.1] | 5.3 [4.8 to 6.2] | 5.1 [4.5 to 7.0] | 8.3 [6.5 to 11.1]

23. Secondary Outcome: Serum Creatine Concentration in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2015
Description: Serum creatine concentration (μmol/L) was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2015. The Arms A, B, C, D - inpatients only were mutually exclusive in 2015.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2015, up to 1 day
Population: as for outcome 2
Measure: Median (Inter-Quartile Range); unit: Micromole per liter (μmol/L)
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015
Number analyzed (Participants) | 14240 | 3345 | 4142 | 2622 | 27863
Micromole per liter (μmol/L) | 70.0 [54.1 to 95.8] | 56.0 [46.0 to 68.0] | 67.0 [54.0 to 87.0] | 62.3 [52.0 to 73.0] | 68.0 [54.1 to 88.0]

24. Secondary Outcome: Serum Creatine Concentration in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2017
Description: Serum creatine concentration (μmol/L) was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2017. The Arms A, B, C, D - inpatients only were mutually exclusive in 2017.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2017, up to 1 day
Population: as for outcome 3
Measure: Median (Inter-Quartile Range); unit: Micromole per liter (μmol/L)
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017
Number analyzed (Participants) | 29249 | 7090 | 7533 | 3737 | 52078
Micromole per liter (μmol/L) | 69.2 [55.0 to 95.0] | 54.0 [45.0 to 65.0] | 68.0 [55.0 to 87.0] | 61.0 [51.0 to 71.6] | 67.0 [54.0 to 87.0]

25. Secondary Outcome: Serum Creatine Concentration in Inpatients and in All Participants (in- and Outpatients) at Their Last Visit in 2019
Description: Serum creatine concentration (μmol/L) was calculated for inpatients grouped by their diagnoses category [Arm A, B, C, D - inpatients only] and for all participants [All in- and outpatients] at their last visit in 2019. The Arms A, B, C, D - inpatients only were mutually exclusive in 2019.
  Patients with risk factors (RF) were patients with diagnosis of CVD, HF, CKD or at high CV risk. Each participant could potentially have multiple diagnoses simultaneously.
  The data presented for this outcome is an retrospective analysis of electronic healthcare records of the Tianjin regional data base. Participants with diagnoses of interest were identified by International Classification of Disease (ICD) code.
Time Frame: Last visit in 2019, up to 1 day
Population: as for outcome 4
Measure: Median (Inter-Quartile Range); unit: Micromole per liter (μmol/L)
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
Number analyzed (Participants) | 77928 | 11062 | 15971 | 4904 | 133527
Micromole per liter (μmol/L) | 70.0 [55.9 to 94.0] | 53.5 [45.0 to 65.0] | 68.1 [55.4 to 86.0] | 62.0 [52.4 to 72.0] | 67.6 [54.0 to 87.3]

ADVERSE EVENTS:
Time Frame: On the last visit (1 day) in 2015, 2017, and 2019 data was retrospectively assessed for the last 12 months in 2015, 2017, and 2019.
Description: This is a retrospective non-interventional study based on electronic healthcare records of the Tianjin regional data base containing the information diagnosis of death. Outcome 14, 15 and 16 show the retrospective analysis of number of patients identified as dead by International Classification of Disease (ICD) code and are also reported here. The arms A, B, C, and D were mutually exclusive in each year but not across years. 'Serious' and 'Other Adverse Events' were not collected.
Arm/Group | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2015 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2015 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - 2015 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2015 | All in- and Outpatients in 2015 = Total in 2015 | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2017 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2017 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2017 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2017 | All in- and Outpatients in 2017 = Total in 2017 | Diabetic Inpatients With Risk Factors (RF) [Arm A Inpatients Only] - in 2019 | Diabetic Inpatients Without RF [Arm B Inpatients Only] - in 2019 | Non-diabetic Inpatients With RF [Arm C Inpatients Only] - in 2019 | Non-diabetic Inpatients Without RF [Arm D Inpatients Only] - in 2019 | All in- and Outpatients in 2019 = Total in 2019
All-Cause Mortality (participants affected / at risk) | 303/84600 | 18/14322 | 94/21682 | 15/6573 | 430/398008 | 504/116799 | 29/22121 | 141/26955 | 30/8908 | 704/580958 | 225/139535 | 8/21549 | 41/28868 | 20/9012 | 294/680438
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2021-06-18): https://cdn.clinicaltrials.gov/large-docs/96/NCT04903496/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT04903496/SAP_001.pdf